CLINICAL TRIAL: NCT03761849
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Phase III Clinical Study to Evaluate the Efficacy and Safety of Intrathecally Administered RO7234292 (RG6042) in Patients With Manifest Huntington's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Intrathecally Administered RO7234292 (RG6042) in Participants With Manifest Huntington's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BN40423; GENERATION HD1 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Huntingtons Disease
Keywords: HD, RG6042, intrathecal, ASO, antisense oligonucleotide
MeSH Terms: conditions — Chorea | interventions — tominersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RO7234292 Q8W (Experimental): RO4234292 is administered intrathecally every 8 weeks.
  Interventions: Drug: RO7234292
- RO7234292 Q16W (Experimental): RO7234292 is administered intrathecally every 16 weeks. Participants in this arm will also receive placebo at alternate weeks to keep the blind.
  Interventions: Drug: RO7234292; Drug: Placebo
- Placebo (Placebo Comparator): Placebo will be administered every 8 weeks by IT injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7234292 — Intrathecal injection
  Other Names: Tominersen
  Arms: RO7234292 Q16W; RO7234292 Q8W
Drug: Placebo — Intrathecal injection
  Arms: Placebo; RO7234292 Q16W

SUMMARY:
This study will evaluate the efficacy, safety, and biomarker effects of RO7234292 (RG6042) compared with placebo in participants with manifest Huntington's disease (HD)

ELIGIBILITY:
Inclusion Criteria:

* Manifest HD diagnosis, defined as a DCL score of 4
* Independence Scale (IS) score >= 70
* Genetically confirmed disease by direct DNA testing with a CAP score >400
* Clinical assessment to ensure individual has intact functional independence at baseline to maintain self-care and core activities of daily living (ADLs).

Exclusion Criteria:

* Any serious medical condition or clinically significant laboratory, or vital sign abnormality or claustrophobia at screening that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of study drug

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (96):
- United States (20):
  - Uab Medicine, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Stanford Univ Medical Center, Palo Alto, California
  - SC3 Research Group, Inc, Pasadena, California
  - University of California Davis Medical System, Sacramento, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Georgetown University; Research Division, Psychiatry, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Dent Neurological Institute, Amherst, New York
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston; McGovern Medical School, Houston, Texas
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - Evergreen Health Care Center, Kirkland, Washington
- Argentina (3):
  - Hospital Ramos Mejía, CABA
  - INEBA, Capital Federal
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
- Australia (3):
  - WESTMEAD HOSPITAL; Deparment of Neurology, Westmead, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital; Department of Neurology, Parkville, Victoria
- Austria (2):
  - Uniklinik fuer Neurologie, Medizinische Universitaet Innsbruck; Department fuer Neurologie, Innsbruck
  - Christian-Doppler-Klinik - Universitätsklinikum; Universitätskliniik für Neurologie, Salzburg
- Canada (6):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of British Columbia Hospital; Division of Neurology, Vancouver, British Columbia
  - True North Clinical Research-Halifax, Halifax, Nova Scotia
  - Centre for Movement Disorders, North YORK, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Centre Hospitalier de l?Université de Montréal (CHUM), Montreal, Quebec
- Centro de Trastornos del Movimiento (CETRAM); CETRAM, Santiago, Chile
- Denmark (2):
  - Aarhus Universitetshospital; Neurologisk Afdeling F, Neurogenetisk Afsnit, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, København Ø
- France (7):
  - CHU Angers, Batiement Larrey 2, Neurologie, Angers
  - Hopital Henri Mondor; Service de Neurologie, Créteil
  - Hopital Roger Salengro Service de Neurologie, Lille
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - Hopital Gui de Chauliac; Neurologie, Montpellier
  - Hôpital Pitié Salpêtrère; Département de Génétique et Cytogénétique, Paris
  - CHU toulouse - Hôpital Purpan; Departement de Neurologie, Toulouse
- Germany (8):
  - Uniklinik RWTH Aachen; Klinik für Neurologie, Aachen
  - Charité - Universitätsmed. Berlin, Klinik für Psychiatrie und Psychotherapie; Abt. Neuropsychiatrie, Berlin
  - St. Josef-Hospital, Neurologische Klinik der Ruhr-Uni; Huntington-Center NRW, Abt. Neurodegeneration, Bochum
  - German Center for Neurodegenerative Diseases (DZNE), Bonn
  - Universitätsklinikum Erlangen, Abteilung Molekulare Neurologie, Erlangen
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Zentrum für Seltene Erkrankungen, Lübeck
  - George-Huntington- Institut GmbH; Technologiepark Münster, Münster
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
- Italy (6):
  - IRCCS Casa Sollievo Della Sofferenza; Unità Ricerca e Cura Huntington e Malattie Rare, San Giovanni Rotondo, Apulia
  - IRCCS Istituto delle Scienze Neurologiche; UOC Clinica Neurologica, Bologna, Emilia-Romagna
  - Azienda Ospedaliera Sant'Andrea; UOC Neurologia, Rome, Lazio
  - Irccs A.O.U.San Martino Ist; Dinogmi, Genoa, Liguria
  - Fondazione IRCCS Istituto Neurologico Carlo Besta; U.O.C. Genetica Medica-Neurogenetica, Milan, Lombardy
  - A.O.U. Careggi; Diaprtimento Scienze Neurologiche e Psichiatriche, Florence, Tuscany
- Japan (5):
  - Kuwana City Medical Center, Mie
  - National Hospital Organization Niigata National Hospital, Niigata
  - Okayama University Graduate School of Medicine, Densitry and Pharmaceutical Sciences., Okayama
  - Osaka General Medical Center, Osaka
  - National Center of Neurology and Psychiatry, Tokyo
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - LUMC, Leiden
- New Zealand (3):
  - Auckland DHB - Neurlogy Department; Neurology Department, Auckland
  - New Zealand Brain Research Institute, Christchurch
  - Wellington Hospital; Department of Neurology, Wellington
- Poland (3):
  - Szpital Sw. Wojciecha; Oddzial Neurologiczny, Gdansk
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii K, Krakow
  - Instytut Psychiatrii i Neurologii, Warsaw
- Russia (3):
  - FSBHI Siberian Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk, Krasnoyarsk Krai
  - Research Center of Neurology; Neurology Department #5, Moskva, Moscow Oblast
  - ?linical hospital at Kazan station, Republican Center for Movement Disorders and Botulinum Therapy, Kazan', Tatarstan Republic
- Spain (9):
  - Hospital de Cruces; Servicio de Neurologia, Barakaldo, Vizcaya
  - Hospital Universitario de Badajoz; Servicio de Neurología, Badajoz
  - Hospital Clinic Servicio de Neurologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Hospital Universitario de Burgos. Servicio de Neurología, Burgos
  - Hospital Ramon y Cajal; Servicio de Neurologia, Madrid
  - Fundacion Jimenez Diaz; Servicio de Neurología, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Neurologia, Seville
  - Hospital Universitario la Fe; Servicio de Neurologia, Valencia
- Switzerland (2):
  - Universitätsspital Basel; Neurologie, Basel
  - Neurozentrum Siloah, Gümligen
- United Kingdom (11):
  - Aberdeen Royal Infirmary; Medical Genectics, Aberdeen
  - Queen Elizabeth Hospital, Birmingham
  - Cambridge Centre for Brain Repair; Department of Clinical Nuerosciences, Addenbrookes Hospital, Cambridge
  - University Hospital of Wales; Division of Psychological Medicine and Clinical Neurosciences, Cardiff
  - Queen Elizabeth University Hospital Glasgow, Glasgow
  - Leeds General Infirmary, Leeds
  - National Hospital For Neurology and Neurosurgery, London
  - Central Manchester University Hospitals NHS Foundation Trust; Manchester Centre for Genomic Medicine, Manchester
  - John Radcliffe Hospital, Oxford
  - Royal Hallamshire Hospital, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southhampton

REFERENCES:
- [Derived] Rodrigues FB, Ferreira JJ, Wild EJ. Huntington's Disease Clinical Trials Corner: June 2019. J Huntingtons Dis. 2019;8(3):363-371. doi: 10.3233/JHD-199003. PMID 31381524
- [Derived] Rodrigues FB, Quinn L, Wild EJ. Huntington's Disease Clinical Trials Corner: January 2019. J Huntingtons Dis. 2019;8(1):115-125. doi: 10.3233/JHD-190001. PMID 30776019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study BN40423 was originally designed (under Protocol v1-3) to include three dosing regimens under a double-blinded monthly dosing paradigm: tominersen Q4W, tominersen every 8 weeks (Q8W) with alternating placebo, and placebo Q4W. The Sponsor decided to stop enrollment into the ODC and NDC started with new participants with 120mg tominersen Q8W and Q16W
Pre-assignment Details: The study has 2 parts: Original Design Cohorts (ODC) and New Design Cohorts. (NDH) Participants in the two parts' cohorts are separate and sequential.
Groups:
- Placebo ODC: Matching Placebo Q4W
- RO7234292 Q4W ODC: RO7234292 120 mg Q4W
- RO7234292 Q8W ODC: RO7234292 120 mg Q8W
- Tomi 120 mg Q8W NDC; Tomi 120mg Q16W NDC; Placebo NDC: NDC Arms were enrolled after the completion of ODC
Period: Overall Study
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Started | 36 | 36 | 36 | 263 (NDC Arms were enrolled after the completion of ODC) | 264 (NDC Arms were enrolled after the completion of ODC) | 264 (NDC Arms were enrolled after the completion of ODC)
Completed (Participants were transferred to Open Label Extension) | 0 | 0 | 0 | 216 | 207 | 211
Not Completed | 36 | 36 | 36 | 47 | 57 | 53
Not completed — transferred to OpenLabelExtension | 35 | 34 | 36 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 41 | 43 | 35
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2 | 4 | 5
Not completed — Repeated MRI dId not pass QC. | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 4 | 4
Not completed — Death | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 2 | 1
Not completed — Participant could not come to site | 0 | 0 | 0 | 0 | 1 | 0
Not completed — SF- safety Finding | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Patient did not attend visit | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ODC and NDC ARE mutually exclusive arms. No patients in ODC were enrolled in NDC
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC | Total
Number analyzed (Participants) | 36 | 35 | 36 | 260 | 261 | 260 | 888
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Not all participants were dosed. ODC and NDC are not mutually exclusive arms. First ODC participants completed the milestone and afterwards, different NDC participants were enrolled
  Years | 45.2 (11.0) | 44.9 (9.8) | 47.7 (9.7) | 47.8 (9.6) | 47.5 (9.3) | 48.7 (9.9) | 47.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all participants were dosed. ODC and NDC are not mutually exclusive arms. First ODC participants completed the milestone and afterwards, different NDC participants were enrolled
  Participants
    Female | 22 | 16 | 23 | 111 | 128 | 113 | 413
    Male | 14 | 19 | 13 | 149 | 133 | 147 | 475
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Evaluable participants data are included
  Participants
    number analyzed (Participants) | 36 | 35 | 36 | 260 | 261 | 259 | 887
    Hispanic or Latino | 8 | 3 | 7 | 34 | 38 | 30 | 120
    Not Hispanic or Latino | 28 | 32 | 29 | 222 | 215 | 222 | 748
    Unknown or Not Reported | 0 | 0 | 0 | 4 | 8 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Asian | 1 | 0 | 0 | 5 | 4 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 0 | 3
  White | 33 | 35 | 36 | 246 | 245 | 246 | 841
  More than one race | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 7 | 8 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Composite Unified Huntington's Disease Rating Scale (cUHDRS) Score-Z Score
Description: cUHDRS includes the Total Functional Capacity (range, 0-13; higher score means better functioning), Total Motor Score (range, 0-124; higher score means worse motor severity), Symbol Digit Modality Test (range, 0-110, correctly paired numbers-symbols in 90 seconds; higher score means better cognitive performance), and Stroop Word Reading (range, 0-no max value, correctly read colour words in 45 seconds; higher score means better cognitive performance) scores. A z-score for each test is calculated, which alone can be used to describe relationship between an individual's test score and the mean score of a target population. A z-score of 0 is the mean, and ±1 is 1 standard deviation from the mean. For cUHDRS, z-scores of each test are summed, whereby a higher cUHDRS score is better (score of -3.06-no max value) and a change of ≥1.2 is a meaningful worsening, shown to track functional decline.
Time Frame: Weeks 21 for ODC and 69 for NDC
Population: ITT Population. Only those participants who contributed to data reported in the table. All other data were not evaluable.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 28 | 29 | 25 | 260 | 261 | 260
Scores on a Scale
  Week 21: number analyzed (Participants) | 28 | 29 | 25 | 0 | 0 | 0
  Week 21 | 0.103 (0.193) | -0.367 (0.189) | -0.139 (0.197) |  |  |
  Week 69: number analyzed (Participants) | 0 | 0 | 0 | 260 | 261 | 260
  Week 69 |  |  |  | -1.173 (0.091) | -0.793 (0.093) | -0.630 (0.091)

2. Primary Outcome: Change From Baseline in the Total Functional Capacity (TFC) Score
Description: Total Functional Capacity (TFC) Scores are reported at Weeks 21 and 69. Total Functional Capacity Score ranges from 0 to 13, with a higher score representing better functioning.
Time Frame: Weeks 21 for ODC and 69 for NDC
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 29 | 30 | 25 | 203 | 199 | 206
Scores on a Scale
  Week 21: number analyzed (Participants) | 29 | 30 | 25 | 0 | 0 | 0
  Week 21 | 0.150 (0.246) | -0.463 (0.242) | -0.460 (0.255) |  |  |
  Week 69: number analyzed (Participants) | 0 | 0 | 0 | 203 | 199 | 206
  Week 69 |  |  |  | -1.284 (0.124) | -0.921 (0.126) | -0.883 (0.124)

3. Secondary Outcome: Change From Baseline in Total Motor Score (TMS)
Description: The TMS score is the sum of the individual motor ratings obtained from administration of the 31-item motor assessment. The score ranges from 0 to 124, with a higher score representing more severe impairment.
Time Frame: Weeks 21 for ODC and 69 for NDC
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 29 | 30 | 25 | 200 | 193 | 203
Score on a Scale
  Week 21: number analyzed (Participants) | 29 | 30 | 25 | 0 | 0 | 0
  Week 21 | -1.977 (1.407) | 2.570 (0.542) | 1.493 (0.78) |  |  |
  Week 69: number analyzed (Participants) | 0 | 0 | 0 | 200 | 193 | 203
  Week 69 |  |  |  | 4.028 (0.575) | 3.524 (0.583) | 3.513 (0.573)

4. Secondary Outcome: Change From Baseline in Symbol Digit Modalities Test (SDMT) Scores' Least Squares Mean Values
Description: Symbol Digit Modality Test -SDMT test measures the number of items correctly paired maximum of 110 correct pairs in 90 seconds, more correctly paired items representing less impairment.
  The differences in LS mean ( +/-SE) change from baseline SDMT score between the active groups compared with the placebo group at Weeks 21 and 69 were reported. A negative change from baseline in the SDMT indicates disease progression.
  The Least Square Mean values of Symbol Digit Modality Test Scores are reported below.
  The minimum range for the SDMT scale is 0, indicating highest severity. A max number is not possible as it is a time based task, based on the number of correct answers within a set time frame. There are no validated SDMT score thresholds to indicate the level of HD symptom severity.
Time Frame: Weeks 21 for ODC and 69 NDC
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 28 | 29 | 27 | 200 | 193 | 202
Scores on a scale
  Week 21: number analyzed (Participants) | 28 | 29 | 27 | 0 | 0 | 0
  Week 21 | 1.865 (0.886) | -1.166 (0.867) | 1.204 (0.879) |  |  |
  Week 69: number analyzed (Participants) | 0 | 0 | 0 | 200 | 193 | 202
  Week 69 |  |  |  | -2.641 (0.380) | -0.996 (0.385) | -0.216 (0.379)

5. Secondary Outcome: Change From Baseline in Stroop Word Reading (SWR) Test Scores' Least Squares Mean Values
Description: Stroop Word Reading-SWR number of words and colors read correctly is counted, with a higher score indicating better cognitive performance scores. There is no upper limit for SWR as it is a time based task. The lower limit (worst possible) however is 0; higher score is better meaning less severity.
  The differences in LS mean ( +/-SE) change from baseline SWR score between the active groups compared with the placebo group at Weeks 21 and 69 were reported. A negative change from baseline in the SWR indicates disease progression.
  The Least Square Mean values of Stroop Word Reading (SWR) Test Scores are reported below.
Time Frame: Weeks 21 for ODC and 69 for NDC
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 28 | 29 | 27 | 200 | 193 | 202
Scores on a Scale
  Week 21: number analyzed (Participants) | 28 | 29 | 27 | 0 | 0 | 0
  Week 21 | -1.397 (1.902) | 0.469 (1.847) | -1.036 (1.842) |  |  |
  Week 69: number analyzed (Participants) | 0 | 0 | 0 | 200 | 193 | 202
  Week 69 |  |  |  | -5.224 (0.803) | -3.949 (0.815) | -2.555 (0.802)

6. Secondary Outcome: Change From Baseline in the Clinical Global Impression, Severity Scale (CGI-S) Scores' Least Squares Mean Values
Description: The CGI-S is a single-item measure of current global severity and is completed by the clinician at specified clinic visits. The CGI-S is assessed using an 11-point numeric rating scale (NRS), where higher scores indicate greater severity. Only NDC participants data were reported, all other data were not available.
  CGI-S) Scores range from 0 (not at all severe) to 10 (Extremely severe); lower score is better meaning less severity.
Time Frame: Week 69 for NDC Only
Population: ITT Population. Only those participants who were contributed data reported in the table. All other data were not evaluable. No data could be reported in ODC Arms due to no data were collected.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 0 | 0 | 0 | 200 | 197 | 203
Scores on a Scale |  |  |  | 0.662 (0.093) | 0.640 (0.094) | 0.545 (0.093)

7. Secondary Outcome: Percentage of Patients With a Decrease From Baseline of >=1 Point on the Total Functional Capacity (TFC) Score
Description: Only NDC participant data are available and reported. Total Functional Capacity-TFC score ranges from 0 to 13, with a higher score representing better functioning.
  In this outcome measure, participants with 1 or higher point score decrease from the Baseline TFC Total Score was considered. The Percentage of these participants with such a change was calculated.
Time Frame: Week 69 for NDC only
Population: ITT Population. Only those participants who contributed to data reported in the table. All other data were not evaluable. No data could be reported in ODC Arms due to no data were collected.
Measure: Number; unit: Percentage
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 0 | 0 | 0 | 260 | 261 | 260
Percentage
  Week 69 Decline from baseline at least 1.2 points Yes |  |  |  | 55.7 | 50.3 | 49.5
  Week 69 Decline from baseline at least 1.2 points No |  |  |  | 44.3 | 49.7 | 43.7

8. Secondary Outcome: Percentage of Patients With a Decline From Baseline of >=1.2 Points on the Composite Unified Huntington's Disease Rating Scale-cUHDRS Score
Description: Only NDC participant data are available and reported. The cUHDRS is comprised of the sum scores of the subscales, score ranges and severities mentioned in the Outcome Measure Description 1 (please see above).
  In this outcome measure, participants with 1.2 or higher point score decrease from the Baseline Composite Unified Huntington's Disease Rating Scale- cUHDRS Total Score was considered. The Percentage of these participants with such a change was calculated.
  cUHDRS lowest (worst) score possible value is -3.06 but no upper limit as it involves SWR; higher score is better meaning less severity.
Time Frame: Week 69 for NDC Only
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 0 | 0 | 0 | 260 | 261 | 260
Percentage of Participants
  Week 69 Yes |  |  |  | 44.5 | 32.1 | 29.7
  Week 69 No |  |  |  | 55.5 | 67.9 | 70.3

9. Secondary Outcome: Percentage of Patients With an Unchanged or Improved Score on the Clinical Global Impression, Change Scale Score
Description: The Clinical Global Impression, Change - CGI-C Scale is a single-item measure of change in global status scale and total scores are summed and reported. The CGI-C has 7 response options: "very much worse," "much worse," "minimally worse," "no change," "minimally improved," "much improved," and "very much improved." "Yes", "No" responses collected and total scores are summed and reported below. Percentage of participants who have unchanged or improved scores from the Baseline CGI-C Scores are calculated and reported here.
  Total CGI-C scores range from 1 (Very much improved) to 7 (Very much worse); lower score is better meaning less severity. Only NDC Arms data were available. Minimum and maximum values are 1 and 7 respectively.
Time Frame: Weeks 53 and 69 NDC only
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 0 | 0 | 0 | 260 | 261 | 260
Percentage of Participants
  Week 69 Yes |  |  |  | 55.4 | 59.6 | 56.3
  Week 69 No |  |  |  | 44.6 | 40.4 | 43.7

10. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Up to 117 Weeks (29 months)
Population: Safety Population
Measure: Number; unit: Percentage
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 36 | 35 | 36 | 260 | 261 | 260
Percentage | 77.8 | 80.0 | 61.1 | 92.3 | 90.0 | 93.1

11. Secondary Outcome: Change From Baseline in Montreal Cognitive Assessment (MoCA)
Description: ODC Week 21 and NDC Week 69 data were reportable. Total MOCA scores are reported. The MoCA is a patient-completed assessment used to detect cognitive impairment. It contains a series of basic assessments, including attention and visuospatial tasks. The total score ranges from 0-30, where lower scores indicate greater impairment.
Time Frame: Up to Week 21 for ODC, Up to Week 69 for NDC
Population: ITT Population. Only those participants who were contributed data reported in the table. All other data were not evaluable.
  NDC participants number are different at Week 21 and 69, reported data are from all evaluable participants.
Measure: Mean (Standard Deviation); unit: Scores on a Sclae
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 28 | 29 | 27 | 250 | 246 | 256
Scores on a Sclae
  Week 21 | -0.07 (0.86) | 0.10 (1.37) | 0.33 (0.92) | 0.44 (2.91) | 0.39 (2.66) | 0.45 (2.29)
  Week 69: number analyzed (Participants) | 0 | 0 | 0 | 234 | 231 | 232
  Week 69 |  |  |  | 0.15 (3.26) | 0.43 (3.22) | 0.61 (2.44)

12. Secondary Outcome: Percentage of Participants With Suicidal Ideation or Behavior, as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: SI-Suicidal Idealation. For ODC, only Treatment Emergent Suicide-Related Events Based on the Columbia-Suicide Severity Rating Scale (CSSRS) are reported. Four constructs are measured: severity of ideation, intensity of ideation, behavior, and lethality of actual suicide attempts. Binary (yes/no) data are collected for 10 categories, and composite endpoints based on the categories are followed over time to monitor patient safety (Posner et al. 2011). It maps to the Columbia-Classification Algorithm for Suicide Assessment and meets the criteria listed in the U.S. FDA draft guidance for assessment of suicidality in clinical trials (FDA 2012). The higher scores indicate higher severity
Time Frame: For ODC at 13th Month, for NDC at Week 101
Population: Safety Population
Measure: Number; unit: Percentage
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 35 | 35 | 35 | 259 | 260 | 260
Percentage
  Suicidal Ideation (1-5) 1) Wish to Be Dead | 0 | 8.6 | 2.8 | 9.7 | 11.2 | 10.4
  Suicidal Ideation (1-5) 2) Non-specific Active Suicidal Thoughts | 0 | 8.6 | 2.8 | 6.9 | 5.8 | 5.8
  SI(1-5) 3) Active Suicidal Ideation with Methods (Not Plan) without Intent to Act | 0 | 2.9 | 0 | 3.5 | 3.5 | 4.2
  Suicidal Ideation (1-5) 4) Active Suicidal Ideation with Some Intent to Act, without Specific Plan | 0 | 0 | 0 | 2.3 | 0.4 | 1.2
  Suicidal Ideation (1-5) 5) Active Suicidal Ideation with Specific Plan and Intent | 0 | 0 | 0 | 1.9 | 0 | 1.2
  Suicidal Behavior (6-10) 6) Preparatory Acts or Behavior | 0 | 0 | 0 | 0.8 | 0.8 | 0.8
  Suicidal Behavior (6-10) 7) Aborted Attempt | 0 | 0 | 0 | 0.4 | 0.4 | 0.4
  Suicidal Behavior (6-10)8)Interrupted Attempt | 0 | 0 | 0 | 0 | 0.4 | 0.4
  Suicidal Behavior (6-10) 9) Non-fatal Suicide Attempt | 0 | 0 | 0 | 1.5 | 1.5 | 1.5
  Suicidal Behavior (6-10) 10) Completed Suicide | 0 | 0 | 0 | 0 | 0 | 0
  Self-injurious Behavior without Suicidal Intent | 0 | 0 | 0 | 0.4 | 1.2 | 1.2
  Suicidal Ideation or Behavior1-5) | 0 | 8.6 | 2.8 | 10.0 | 11.2 | 10.8

13. Secondary Outcome: Concentration of RO7234292 in Plasma
Description: Concentration of tominersen in plasma reported
Time Frame: Week 21 for ODC and Week 69 for NDC
Population: Pharmacokinetic Population. Only those participants who were contributed data reported in the table. All other data were not evaluable.
  NDC participants number are different at Week 21 and 69, reported data are from all evaluable participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 0 | 35 | 36 | 250 | 243 | 0
ng/mL
  Week 21 Pre--dose |  | 0.511 (0.523) | 0.203 (0.0948) | 0.20 (0.37) | 0.06 (0.22) |
  Week 69 Pre dose: number analyzed (Participants) | 0 | 0 | 0 | 214 | 200 | 0
  Week 69 Pre dose |  |  |  | 1.63 (3.40) | 0.28 (0.75) |

14. Secondary Outcome: Trough Concentration of RO7234292 in Cerebrospinal Fluid (CSF)
Description: Tominersen concentrations in cerebrospinal fluid
Time Frame: Week 21 for ODC and Week 69 for NDC
Population: as for outcome 13
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 0 | 35 | 36 | 189 | 182 | 0
ng/mL
  Week 21: number analyzed (Participants) | 0 | 35 | 36 | 149 | 142 | 0
  Week 21 |  | 4.44 (2.24) | 1.51 (0.604) | 1.54 (0.99) | 0.70 (2.29) |
  Week 69: number analyzed (Participants) | 0 | 0 | 0 | 189 | 182 | 0
  Week 69 |  |  |  | 1.74 (1.08) | 0.55 (2.43) |

15. Secondary Outcome: Incidence of Anti-Drug Antibodies (ADAs).
Description: Data at Weeks 21 and 69 for Old Design and New Design Cohorts are reported respectively. All other timepoints were not evaluable and not meaningful.
Time Frame: Week 21 for ODC and Week 69 for NDC
Population: Pharmacokinetic Population. Only those participants who were contributed data reported in the table. All other data were not evaluable.
Measure: Number; unit: Percentage
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 0 | 29 | 27 | 190 | 261 | 260
Percentage
  Week 21 Total Negative: number analyzed (Participants) | 0 | 29 | 27 | 0 | 0 | 0
  Week 21 Total Negative |  | 94.3 | 91.7 |  |  |
  Week 21 Negative Treatment All Samples: number analyzed (Participants) | 0 | 29 | 27 | 0 | 0 | 0
  Week 21 Negative Treatment All Samples |  | 91.4 | 91.7 |  |  |
  Week 21 Total Positive Treatment unaffected: number analyzed (Participants) | 0 | 29 | 27 | 0 | 0 | 0
  Week 21 Total Positive Treatment unaffected |  | 2.9 | 0 |  |  |
  Week 69 Total Negative: number analyzed (Participants) | 0 | 0 | 0 | 190 | 186 | 12
  Week 69 Total Negative |  |  |  | 71.1 | 81.7 | 100
  Week 69 Negative Treatment Unaffected: number analyzed (Participants) | 0 | 0 | 0 | 190 | 186 | 12
  Week 69 Negative Treatment Unaffected |  |  |  | 0 | 1.1 | 0.5
  Week 69 Total Positive: number analyzed (Participants) | 0 | 0 | 0 | 190 | 186 | 12
  Week 69 Total Positive |  |  |  | 28.9 | 18.3 | 22.0
  Week 69 Positive Treatment Induced: number analyzed (Participants) | 0 | 0 | 0 | 190 | 261 | 260
  Week 69 Positive Treatment Induced |  |  |  | 0 | 0 | 0

16. Secondary Outcome: Titer and Antibody Subtype, Determined if ADAs Are Identified
Description: Titer and Antibody Subtype was not analyzed and there is not data to report due to participants' discontinuation
Time Frame: Week 21 for ODC and Week 69 for NDC
Population: No participants and no data to report
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in CSF mHTT Protein Level
Description: Data to be reported within 12 months after the primary completion.
Time Frame: Baseline, Week 101
Reporting Status: Not Posted, anticipated posting 2024-03

18. Secondary Outcome: Change From Baseline in Whole and Regional Brain Volumes, as Detrmined by Structural Magnetic Resonance Imaging (MRI)
Description: Data reported only for ODC Arms. Analysis of Percent Change from Baseline in Volumetric MRI / BSI at 3 Months reported. Analysis performed using analysis of covariance with covariates of CAP, CAG, Age at Baseline and treatment included.
  Analysis of Change from Baseline in: Caudate Volume (mL)
Time Frame: Week 13 for ODC
Population: Pharmacokinetic Population. Only those participants who were contributed data reported in the table. All other data were not evaluable. No data could be reported in NDC Arm Week due to no data were collected, no participants were involved in this Arm.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 34 | 31 | 32 | 0 | 0 | 0
mL
  Week 13 Analysis of Change from Baseline in: Caudate Volume (mL): number analyzed (Participants) | 30 | 24 | 27 | 0 | 0 | 0
  Week 13 Analysis of Change from Baseline in: Caudate Volume (mL) | 0.996 (0.444) | 0.330 (0.491) | 1.124 (0.467) |  |  |
  Week 13 Change from Baseline in: Ventricle Volume (mL) | 1.537 (0.686) | 3.785 (0.718) | 2.011 (0.700) |  |  |
  Week 13 Change from Baseline in: Whole Brain Volume (mL): number analyzed (Participants) | 31 | 30 | 30 | 0 | 0 | 0
  Week 13 Change from Baseline in: Whole Brain Volume (mL) | 0.189 (0.119) | -0.184 (0.123) | -0.133 (0.121) |  |  |

19. Secondary Outcome: Change From Baseline in CSF Neurofilament Light Chain (NfL) Proteint Level
Time Frame: Week 21 for ODC, Weeks 21 and 69 for NDC
Population: ITT Population. Only those participants who were contributed data reported in the table. All other data were not evaluable. No data could be reported in ODC Arm Week 69 due to no data were collected.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Placebo ODC | RO7234292 Q4W ODC | RO7234292 Q8W ODC | Tomi 120 mg Q8W NDC | Tomi 120mg Q16W NDC | Placebo NDC
Number analyzed (Participants) | 28 | 28 | 27 | 224 | 209 | 225
ng/mL
  Week 21 | 12.233 [0.729 to 25.050] | 34.548 [20.671 to 50.022] | 16.553 [4.497 to 29.999] | 31.893 [24.946 to 39.226] | 5.406 [-0.335 to 11.479] | 3.365 [-2.077 to 9.109]
  Week 69: number analyzed (Participants) | 0 | 0 | 0 | 172 | 163 | 169
  Week 69 |  |  |  | 9.996 [3.538 to 16.858] | -2.559 [-8.439 to 3.699] | 5.982 [-0.293 to 12.652]

ADVERSE EVENTS:
Time Frame: For ODC Up to 13 Months. For NDC Approximately Up to 137 Weeks
Groups:
- PLB ODC: Placebo Q4W every 16 Week
- Q4W ODC: RO7234292 loading dose: 120 mg at every 16 Week
- Q8W ODC: RO7234292: 120 mg Q8W from Week 1 to Week 69
- Q8W NDC; Q16W NDC; PLB NDC: NDC Arms were enrolled after the completion of ODC
Arm/Group | PLB ODC | Q4W ODC | Q8W ODC | Q8W NDC | Q16W NDC | PLB NDC
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 1/263 | 2/264 | 3/264
Serious Adverse Events (participants affected / at risk) | 2/36 | 1/36 | 1/36 | 50/263 | 28/264 | 34/264
Other Adverse Events (participants affected / at risk) | 24/36 | 23/36 | 19/36 | 204/263 | 187/264 | 193/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLB ODC (N=36) | Q4W ODC (N=36) | Q8W ODC (N=36) | Q8W NDC (N=263) | Q16W NDC (N=264) | PLB NDC (N=264)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Wound haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Water intoxication (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chorea (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Demyelination (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Assisted suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusion of parasitosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, tactile (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impulse-control disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Persecutory delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 3 (3)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subclavian artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLB ODC (N=36) | Q4W ODC (N=36) | Q8W ODC (N=36) | Q8W NDC (N=263) | Q16W NDC (N=264) | PLB NDC (N=264)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2) | 17 (20) | 15 (16) | 19 (20)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 12 (14) | 12 (17) | 15 (19)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 14 (17) | 16 (22) | 16 (20)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 10 (13) | 17 (20) | 10 (10)
Gait disturbance (General disorders) | 0 (0) | 4 (4) | 1 (2) | 10 (11) | 3 (3) | 2 (2)
Puncture site pain (General disorders) | 0 (0) | 2 (3) | 2 (2) | 24 (45) | 13 (17) | 24 (46)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (2) | 12 (13) | 14 (17) | 13 (16)
Fungal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 36 (48) | 28 (40) | 44 (61)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (5) | 2 (2) | 13 (20) | 13 (14) | 8 (18)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 16 (19) | 15 (20) | 18 (30)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 2 (2) | 4 (6) | 70 (136) | 63 (141) | 79 (170)
Inappropriate schedule of product administration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 1 (2)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 4 (6) | 3 (6) | 7 (8) | 24 (34) | 18 (28) | 21 (39)
Procedural pain (Injury, poisoning and procedural complications) | 4 (8) | 6 (11) | 5 (9) | 23 (51) | 21 (31) | 22 (29)
CSF protein increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 13 (13) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 19 (22) | 12 (13) | 22 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2) | 4 (4) | 57 (91) | 58 (93) | 49 (92)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 19 (30) | 14 (16) | 15 (20)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0) | 1 (1) | 20 (33) | 22 (31) | 17 (19)
Headache (Nervous system disorders) | 6 (9) | 3 (3) | 4 (6) | 61 (150) | 57 (105) | 59 (114)
Paraesthesia (Nervous system disorders) | 3 (4) | 2 (2) | 2 (4) | 7 (10) | 8 (10) | 6 (10)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 10 (15) | 4 (4) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 16 (20) | 11 (12) | 15 (16)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 11 (14) | 15 (16) | 13 (16)
Skin laceration (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 12 (14) | 5 (5) | 8 (11)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (5) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT03761849/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT03761849/SAP_001.pdf